CLINICAL TRIAL: NCT04843826
Title: تعديل النسيج الضام عنيق تحت الظهارة من أجل إعادة بناء حليمي بين الأسنان حول الزراعه المتأخره في المنطقة الجمالية
Brief Title: Modified Pedicle Subepithelial Connective Tissue Graft for Interdental Papillary Reconstruction Around Delayed Implants in the Esthetic Zone: A Case Series Trail
Acronym: delay implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Sadek Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ahmed Sadek Mohamed, teacher assistance, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER 111; per 122 (Registry Identifier: implant)
Record Dates: First submitted 2021-04-04; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-04

CONDITIONS: Papilla Reconstruction

STUDY DESIGN:
Intervention Model Description: Case Series trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- delayed implant (Experimental): 1. Patients 18 years or older.
  2. Periodontally and systemically healthy.
  3. Sufficient bone width and height for implant placement
  4. Adequate mesiodistal width and inter-arch space for placement of a delayed implant.
  5. Full mouth plaque index less than 15% (Bentley and Disney, 1995)
  6. cooperative patients who will comply to follow up visits
  Interventions: Procedure: papilla reconstruction

INTERVENTIONS:
Procedure: papilla reconstruction — subepithelial connective tissue graft for interdental papillary reconstruction around delayed
  Other Names: create papilla around delayed implant

SUMMARY:
This case series trial aims to evaluate the effect of a modified pedicle subepithelial connective tissue graft in creating anatomical papilla around one-stage delayed implant in the esthetic zone to establish better esthetics.

DETAILED DESCRIPTION:
* Preparation of the implant site will be prepared by a crestal incision on the ridge bisecting the existing keratinized mucosa and vertical releasing incisions extending to the vestibule. The papillae of the adjacent teeth are not included in the flap design.
* A full thickness flap will be raised buccally exposing the underlined ridge of the implant site. A surgical drill guide will be used for the precise placement of the pilot drill. After pilot drill application, the osteotomy will be prepared with the corresponding size of parallel drill.
* The implant will be placed in the recipient site by means of an insertion device. The implant neck will be positioned flushing with the crestal bone level.
* The healing abutment extension of the implant will be placed in such a way that the head of the implant protruded about 2 to 3 mm from the bone crest.
* Reassessment of the case to assure absence of any signs of inflammation and presence of normal tissues before the surgical procedure

ELIGIBILITY:
Exclusion Criteria:

1. Pregnant females.
2. Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, et al., 2009)
3. Handicapped and mentally retarded patients.
4. Patients undergoing radiotherapy.
5. Presence of systemic disease that would affect wound healing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-09-14 (Estimated)

PRIMARY OUTCOMES:
papilla height | 3 month
  Periodontal probe and reference line

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No